CLINICAL TRIAL: NCT00969137
Title: Sensitivity to Intravenous Nicotine: Genetic Moderators
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Mehmet Sofuoglu, Principle Investigator, Yale University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 0905005103; R03DA027474 (NIH); DCNBR / CNB (Other: NIDA)
Record Dates: First submitted 2009-08-31; First posted 2009-09-01 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Nicotine Dependence
Keywords: smoking, nicotine, cigarettes
MeSH Terms: conditions — Tobacco Use Disorder; Smoking | interventions — Sodium Chloride; Nicotine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nicotine (Active Comparator): Intravenous Nicotine
  Interventions: Drug: Nicotine
- Saline (Placebo Comparator): Saline infusion
  Interventions: Drug: saline

INTERVENTIONS:
Drug: saline — intravenous saline
  Arms: Saline
Drug: Nicotine — Intravenous nicotine
  Arms: Nicotine

SUMMARY:
To determine if the mu opioid receptor gene (OPRM1) A118G polymorphism moderates the subjective-rewarding effects of intravenous (IV) nicotine in male and female smokers. The subjective effects of nicotine will be measured with a Drug Effects Questionnaire, including the ratings of "good effects" and "drug liking". We hypothesize that smokers with the AG/GG genotype for the OPRM1 A118G will have attenuated subjective-rewarding effects from IV nicotine when compared to those with AA genotype.

DETAILED DESCRIPTION:
Increasing evidence suggest that MOR contribute to nicotine's rewarding effect. Further, the functional OPRM1 A118G variant has been linked to rewarding effects of alcohol in alcohol users and to nicotine in female smokers. Since no previous studies examined the influence of the A118G variation on pure nicotine responses, the next logical step is to evaluate how this genetic polymorphism affects nicotine's rewarding, cognitive, and physiological effects using IV nicotine administration in male and female smokers. In addition, the association of the G398A polymorphism of the CHRNA5 gene (rs16969968) with maximal response to nicotinic agonists justifies examination of this SNP as a moderator of IV nicotine sensitivity in humans (Bierut et al. 2008). This SNP will be examined in an exploratory fashion since it is not feasible to fully stratify the study sample for multiple SNPs. The frequency of rs16969968 SNP ranges from 35%-42% among those of European ancestry, making it feasible to examine this variation in our subject sample.

Currently this study is active and enrollment is continuing. Currently there are 205 completers and on going.(June 2014)

ELIGIBILITY:
Inclusion Criteria:

* Female and male smokers, aged 18 to 50 years;
* History of smoking daily for the past 12 months, 10-25 cigarettes daily;
* Not seeking treatment at the time of the study for nicotine dependence;
* Have a FTND score of at least 5 and CO level > 10ppm;
* In good health as verified by medical history, screening examination, and screening laboratory tests;
* For women, not pregnant as determined by pregnancy screening, nor breast feeding, and using acceptable birth control methods.

Exclusion Criteria:

* History of major medical illnesses that the physician investigator deems as contraindicated for the patient to be in the study;
* Regular use of psychotropic medication (antidepressants, antipsychotics, or anxiolytics) and recent psychiatric diagnosis and treatment for Axis I disorders including major depression, bipolar affective disorder, schizophrenia or panic disorder;
* Abuse of alcohol or any other recreational or prescription drugs.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 213 (Actual)
Dates: Start 2009-06-02 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
primary hypotheses will test the influence of OPRM1 A118G status on subjective responses to IV nicotine, which will be measured with the drug effects questionnaire (DEQ). | Injections 30 minutes apart

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Sofuoglu, M.D,Ph.D., Principal Investigator — Yale University
Locations (1):
- Department of Veterans Affairs, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No